CLINICAL TRIAL: NCT05757583
Title: Impact of Metabolic Dysfunction and Mucus Plugging on Asthma Physiology
Acronym: IMAP
Status: Recruiting | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 22-37338; R01HL164787 (NIH)
Record Dates: First submitted 2023-02-23; First posted 2023-03-07 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Samples of plasma and serum will be banked in the UCSF Airway Tissue Bank.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Patients with asthma, obesity and metabolic dysfunction: Otherwise healthy asthmatic subjects with:
  1. Body Mass Index (BMI) ≥ 30; and
  2. Metabolic dysfunction evidenced by at least one of the following:
     * high plasma IL-6 (> 3.0 pg/mL)
     * insulin resistance (HOMA-IR > 3 mass units)
- Patients with asthma, obesity and no metabolic dysfunction: Otherwise healthy asthmatic subjects with:
  1. Body Mass Index (BMI) ≥ 30; and
  2. No evidence of metabolic dysfunction
- Patients with severe asthma and mucus plugs: Otherwise healthy asthmatic subjects:
  1. Requiring treatment with high dose inhaled corticosteroids plus a second controller, systemic corticosteroid, or biologic therapy; and
  2. Evidence of mucus plugs as defined by a mucus plug score ≥ 4
- Patients with severe asthma and no mucus plugs: Otherwise healthy asthmatic subjects:
  1. Requiring treatment with high dose inhaled corticosteroids plus a second controller, systemic corticosteroid, or biologic therapy; and
  2. No evidence of mucus plugs as defined by a mucus plug score < 4

SUMMARY:
This is a single-center study of 80 subjects with asthma including those with obesity and metabolic dysfunction (MD), those with obesity and without metabolic dysfunction, those with severe asthma and mucus plugging and those with severe asthma and without mucus plugging. Screening data will be reviewed to determine participant eligibility. Participants who meet all inclusion criteria will participate in a cardiopulmonary exercise testing (CPET) visit to compare lung function markers and change in oxygen saturation between obese patients with and without MD and severe asthma patients with and without mucus plugging.

DETAILED DESCRIPTION:
The mechanism of poor exercise tolerance in patients with severe asthma is poorly understood. In preliminary data, the investigators have identified increases in air trapping in patients with obese asthma and metabolic dysfunction and patients with asthma and mucus plugs. The investigators have also found air trapping on CT (Computerized Tomography) scans of severe asthma patients with mucus plugs. Therefore, the investigators hypothesize that obese patients with metabolic dysfunction (MD) and severe asthma patients with mucus plugs develop changes in lung function during exercise.

To test this hypothesis, this protocol will plan for cardiopulmonary exercise testing in patients with obesity or severe asthma. The analyses will compare dynamic hyperinflation, expiratory flow limitation, and the RV/TLC ratio (ratio of residual volume to total lung capacity) before and after exercise between obese patients with and without MD and severe asthma patients with and without mucus plugs.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥ 18 years old at Visit 0
2. Written informed consent obtained from subject and ability for subject to comply with the requirements of the study.
3. History of physician diagnosed asthma
4. Evidence of bronchodilator reversibility (12% improvement in FEV1 after albuterol administration) or positive methacholine challenge PC20 or PD20. Historical evidence is accepted.
5. Meets criteria for obesity or severe asthma a. Obesity: BMI≥30 i. Metabolic dysfunction is defined as presence of either:

1. IL-6 high: Plasma IL-6 > 3.0 pg/mL 2. Insulin resistance: HOMA-IR > 3 mass units b. Severe asthma: Requires treatment with high dose inhaled corticosteroids plus a second controller, systemic corticosteroid, or biologic therapy.

i. Mucus Plugging is defined as mucus plug score ≥ 4

Exclusion Criteria:

1. Asthma exacerbation or URI within the previous 6 weeks.
2. History of smoking

   1. If <30 years old: Smoked for ≥5 pack-years
   2. If ≥30: Smoked for ≥10 pack years
3. Pregnancy
4. Absolute or relative contraindication to exercise testing per ATS criteria
5. Any other criteria that place the subject at unnecessary risk according to the judgment of the Principal Investigator and/or attending physician of record.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will recruit up to 80 asthma participants, at least 20 with obesity and MD, 20 with obesity and no MD, 20 with severe asthma and mucus plugs and 20 with severe asthma and no mucus plugs.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2023-04-05 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Change in EELV (End Expiratory Lung Volume) | At CPET visit.
  We will compare change in EELV during the CPET (Cardiopulmonary Exercise Test) between the obese asthma patients with MD or without MD and between the patients with severe asthma with mucus plugs or without mucus plugs.

SECONDARY OUTCOMES:
Change in RV (Residual Volume) and TLC (Total Lung Capacity) | At CPET Visit
  We will compare change in RV and TLC during the CPET between the obese asthma patients with MD or without MD and between the patients with severe asthma with mucus plugs or without mucus plugs.
Change in oxygen saturation during exercise | At CPET Visit
  Change in oxygen saturation during the CPET will be assessed and compared between the obese asthma patients with MD or without MD and between the patients with severe asthma with mucus plugs or without mucus plugs.

CONTACTS AND LOCATIONS:
Overall Officials: John Fahy, MD, MS, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF Airway Clinical Research Center, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No